CLINICAL TRIAL: NCT00547508
Title: A Randomized, Double-Blind, Parallel, Placebo-Controlled Study in Men With Erectile Dysfunction to Evaluate the Efficacy and Safety of Tadalafil When Sexual Attempts Occur at Specific Time Points After Dosing
Brief Title: To Determine How Different Doses of Tadalafil Work on Getting and Keeping an Erection 26 or 36 Hours After Taking
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7004; H6D-MC-LVFD
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- 3 (Active Comparator): tadalafil
  Interventions: Drug: tadalafil
- 4 (Active Comparator): tadalafil
  Interventions: Drug: tadalafil
- 5 (Active Comparator): tadalafil
  Interventions: Drug: tadalafil
- 6 (Active Comparator): tadalafil
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — 10 mg tablet taken orally, no more than once a day, at anytime during the 2-4 week equilibration phase and then 24 hours prior to sexual intercourse for 4-6 weeks in the assessment phase
  Other Names: LY450190; Cialis; IC351
  Arms: 4
Drug: placebo — Placebo tablet taken by mouth, no more than once a day, anytime during the 2-4 week equilibration phase and then 24 hours prior to sexual intercourse for 4-6 weeks in the assessment phase
  Arms: 1
Drug: tadalafil — 20 mg tablet taken orally, no more than once a day, at anytime during the 2-4 week equilibration phase and then 24 hours prior to sexual intercourse for 4-6 weeks in the assessment phase
  Other Names: LY450190; Cialis; IC351
  Arms: 5
Drug: tadalafil — 20 mg tablet taken orally, no more than once a day, at anytime during the 2-4 week equilibration phase and then 36 hours prior to sexual intercourse for 4-6 weeks in the assessment phase
  Other Names: LY450190; Cialis; IC351
  Arms: 6
Drug: tadalafil — 10 mg tablet taken orally, no more than once a day, at anytime during the 2-4 week equilibration phase and then 36 hours prior to sexual intercourse for 4-6 weeks in the assessment phase
  Other Names: LY450190; Cialis; IC351
  Arms: 3
Drug: placebo — Placebo tablet taken by mouth, no more than once a day, anytime during the 2-4 week equilibration phase and then 36 hours prior to sexual intercourse for 4-6 weeks in the assessment phase
  Arms: 2

SUMMARY:
Study to see how effective different doses of tadalafil are for getting and keeping an erection when sex is attempted after a certain number of hours.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months history of erectile dysfunction (ED)
* Anticipate a monogamous relationship with a female sexual partner
* Be able to make minimum required sexual intercourse attempts
* Abstain from using any other ED treatment

Exclusion Criteria:

* History of other primary sexual disorder
* Treatment with nitrates
* Have a penile implant or clinically significant penile deformity
* History of certain heart problems
* Do not meet certain lab value reference ranges

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2002-10; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Prove superiority to placebo by measuring question 3 of the SEP diary | 6-10 and 24 weeks

SECONDARY OUTCOMES:
Compare effectiveness when patient can freely choose time of sex versus when time of sex attempt is set by the score of question 3 in the SEP diary | 6-10 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com